CLINICAL TRIAL: NCT06102954
Title: Steps to Avoid Falls in the Elderly- A TECHnology Enhanced Intervention
Brief Title: A Multi-domain and Multi-component Falls Intervention Program for Community- Dwelling Older Adults: SAFE-TECH
Acronym: SAFE-TECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, David Bruce Matchar, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-496
Record Dates: First submitted 2023-10-15; First posted 2023-10-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fall Prevention; Fall Injury
Keywords: Fall; Injurious fall; Falls Prevention Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 12-weeks active intervention session includes exercise and educational components.
  9 months maintenance phase
  Interventions: Other: Falls prevention intervention including exercise and educational components
- Control group (No Intervention): No intervention for 12 months during intervention period.

INTERVENTIONS:
Other: Falls prevention intervention including exercise and educational components — This includes five domains of exercise (strength, balance, flexibility, coordination, and endurance) and educational components to manage other falls risk factors (polypharmacy, nutrition, pain, orthostatic hypotension, poor vision and environmental hazard evaluations).
  Arms: Intervention group

SUMMARY:
Background: Falls and fall-related injuries among older adults are a significant health problem that results in injuries, prolonged hospitalisation, reduced mobility, and poorer quality of life. Previous falls prevention programs have demonstrated the effectiveness of multi-component falls prevention interventions in improving functional outcomes and reducing falls compared to usual care. A previous trial of a tailored multi-component falls intervention program for older adults recruited from the emergency department (SAFE) found that there is significant heterogeneity in terms of falls risk factors in high falls risk older adults. Thus, the effectiveness of SAFE in participants with poorer cognitive function or had more comorbidities were less effective and less cost-effective. Therefore, the aim of this trial is to demonstrate the effectiveness of a technology-enhanced, multi-domain and multi-component falls prevention intervention in reducing number of fallers and injurious fallers among older adults with elevated fall risk.

Hypothesis: Using novel wearable technologies to a) identify older adults who are at high risk of falls and more likely to benefit from a multi-component intervention and b) tailor the exercise and educational components by giving individualized biofeedback will improve the effectiveness of an enhanced multi-domain, multi-component falls intervention program for community dwelling older adults.

Methodology: This study is a randomized controlled trial aimed at demonstrating the effectiveness of a technology-enhanced, multi-domain and multi-component falls prevention intervention (SAFE-TECH) in community- dwelling older adults with elevated fall risk compared with usual care. Participants in both arms are selected based on questionnaire based and wearable sensor based predictions of their falls risk. Participants in the intervention arm will receive a 12-week active falls intervention program consisting of exercise and educational components, with detailed biofeedback of their functional status.

DETAILED DESCRIPTION:
Objective: To demonstrate the feasibility and effectiveness of a technology-enhanced multi-domain, multi-component falls intervention program consisting of screening, assessments, progressive physical therapy and education to reduce falls and injurious falls in community-dwelling older adults in Singapore.

Methodology: This study is a multi-center, two-arm, parallel group, randomized controlled trial with 400 participants allocated to the intervention and control arm in a 1:1 ratio. In the intervention arm, participants will be enrolled in a multi-domain, multi-component falls intervention program that consists of exercise and educational components for 12 weeks. The exercise components are progressive and tailored to individual falls risk factors. Exercises aim to improve 5 domains of physical function: strength, balance, flexibility, coordination, and aerobic endurance. The educational components focus on the management of fall risk factors such as polypharmacy, nutrition, pain, orthostatic hypotension, poor vision, and environmental hazards. The education sessions also provide feedback based on individualized falls risk assessments. After the 12-week active intervention phase, the participants in the intervention arm will enter a 9-month maintenance phase where they will be encouraged to maintain their physical activity, and continue practicing falls prevention behavior.

The study will collect information from both intervention and control arm on their living situation, cognitive function, quality of life, general health, falls history, behavioral and psychosocial characteristics, handgrip strength, orthostatic hypotension, ankle mobility, physical function (Short Performance Physical Battery) and gait assessment (ZurichMOVE system of wearable gait sensors) at baseline, 3rd-months and 12th-months into the study. Monthly follow-up calls will be done to collect participants' fall status, healthcare utilisation, physical activity, and exercise self- efficacy over the 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 95 years
* Ambulatory with or without walking aid
* Does not possess cognitive impairment with an Abbreviated Mental Score-Singapore >=6

Exclusion Criteria:

* Had any significant morbidity:

  * Congestive Heart Failure in the past 6 months
  * Myocardial Infarction in the past 6 months
  * Stroke (Intra-Cranial Haemorrhage) in the past 6 months
  * Concussion or Head Injury in the past 6 months
  * End Stage Renal Failure requiring dialysis
  * Severe Asthma or Chronic Obstructive Pulmonary Disease (COPD) (e.g. Chronic Lung Disease or Chronic Bronchitis or Emphysema), experiencing symptoms at rest or with mild activity
  * Lower Limb Fractures in the past 6 months
* Blindness, with or without the use of any visual aids
* Deafness, with or without the use of any hearing aids
* Currently experiencing one of the following:

  * Chest discomfort, or
  * Breathlessness, or
  * Dizziness, or
  * Profuse sweating
* Had an amputation of any part of the lower limbs except toes, or had an amputation of any toes in the last 30 days
* Currently in a long-term institution
* Currently participating in any randomized clinical or controlled trial that involves physical exercise
* Unwilling to complete the baseline gait assessment, or complete less than 3 minutes of the 5-minute baseline gait assessment

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Fallers | Baseline, Monthly phone call follow-up for 1 year, 12th-month after first intervention session
  Evaluation of number of falls in 12 months

SECONDARY OUTCOMES:
Number of Injurious Fallers | Baseline, Monthly phone call follow-up for 1 year, 12th-month after first intervention session
  Evaluation of number of injurious falls in 12 months
Physical Function | Baseline, 3rd-month and 12th-month after first intervention session
  Evaluation of change in physical function using Short Physical Performance Battery test (SPPB) [range from 0 to 12 score].A higher score represents a higher physical function level.
Fear of Falling | Baseline, 3rd-month and 12th-month after first intervention session
  Evaluation of change in falls efficacy using Iconographical Falls Efficacy Scale (Icon-FES). A higher value represents a high concern for falling.
Practice of Falls Prevention Behaviours | Baseline, 3rd-month and 12th-month after first intervention session
  Evaluation of change in practice of falls prevention behaviours by using Falls Behavioral Scale (FaB). A higher value represents a better practice of falls prevention behaviours.

CONTACTS AND LOCATIONS:
Overall Officials: Matchar David Bruce, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Centre for Ageing Research & Education, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matchar DB, Eom K, Duncan PW, Lee M, Sim R, Sivapragasam NR, Lien CT, Ong MEH. A Cost-Effectiveness Analysis of a Randomized Control Trial of a Tailored, Multifactorial Program to Prevent Falls Among the Community-Dwelling Elderly. Arch Phys Med Rehabil. 2019 Jan;100(1):1-8. doi: 10.1016/j.apmr.2018.07.434. Epub 2018 Aug 27. PMID 30165053
- [Background] Matchar DB, Duncan PW, Lien CT, Ong MEH, Lee M, Gao F, Sim R, Eom K. Randomized Controlled Trial of Screening, Risk Modification, and Physical Therapy to Prevent Falls Among the Elderly Recently Discharged From the Emergency Department to the Community: The Steps to Avoid Falls in the Elderly Study. Arch Phys Med Rehabil. 2017 Jun;98(6):1086-1096. doi: 10.1016/j.apmr.2017.01.014. Epub 2017 Feb 12. PMID 28202383
- [Derived] Lai WX, Koh V, Goh JW, Tan KY, Tan KZ, Pai SGS, Taylor WR, Visaria A, Singh NB, Chan AWM, Matchar DB. Steps to Avoid Falls in the Elderly - a TECHnology Enhanced Intervention (SAFE-TECH) study: randomized controlled trial protocol for a community-based, multi-component fall prevention program. BMC Public Health. 2024 Dec 18;24(1):3464. doi: 10.1186/s12889-024-20947-2. PMID 39695436